CLINICAL TRIAL: NCT00005692
Title: Inflammation Markers Over Time in Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4222; R01HL046696 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2005-03

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Thrombosis; Inflammation
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Thrombosis; Inflammation

SUMMARY:
To determine inflammation markers over time in cardiovascular disease. To test the hypothesis that measures of coagulation and fibrinolysis correlate with the incidence of coronary heart disease (CHD) and other thrombosis related disorders, and to help identify those individuals at greatest risk, using the Cardiovascular Health Study (CHS) and Honolulu Heart Program (HHP) populations. These two genetically distinct populations had different event rates for CHD, and offered a unique opportunity to test associations that were uncovered by comparing results across populations.

DETAILED DESCRIPTION:
BACKGROUND:

Coronary heart disease (CHD) and other thrombosis related disorders are a major source of morbidity and mortality in the United States and the world. To a certain extent they are diseases of the elderly, with the majority of overt CHD occurring in persons over the age of 65. Recently, fibrinogen and factor VII have been implicated as independent CHD risk factors in middle age populations, although causative roles have not been established. These studies increased understanding of the relationship of thrombosis to cardiovascular risk.

DESIGN NARRATIVE:

Beginning in 1992, the study tested the hypothesis that measures of coagulation and fibrinolysis correlated with the incidence of coronary heart disease (CHD) and other thrombosis related disorders, and identified those individuals at greatest risk, using the Cardiovascular Health Study (CHS) and Honolulu Heart Program (HHP) populations. These two genetically distinct populations had different event rates for CHD, and offered a unique opportunity to test associations that were uncovered by comparing results across populations. The study examined selected measures of coagulation and fibrinolysis in individuals 65 years and older: measures of pro-coagulation (factor antigen VII, prothrombin fragment 1.2, fibrinopeptide A and thrombin - antithrombin III complex), measures of coagulation inhibition (protein C and protein S, antithrombin III, and the lipoprotein associated coagulation inhibitor (LACI), and measures of fibrinolysis (plasminogen activator inhibitor-1 (PAI-1), tissue plasminogen activator-PAI-1 complex, plasmin-alpha-2 antiplasmin complex, and Lp(a).

A case/control design was used to determine the relationship between the above measurements and the incidence of CHD (and other thrombosis related disorders). The short and medium term biological variability of the above measures was determined to aid in interpretation of observed differences. Finally, the distribution of the above measurements was established in both cohorts and their relationships to other variables in the extensive CHS and HHP data bases ascertained.

The study was renewed in 1999 to determine inflammation markers over time in cardiovascular disease.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Dates: Start 1992-04; Study Completion 2002-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell Tracy — University of Vermont

REFERENCES:
- [Background] Tracy RP, Lemaitre RN, Psaty BM, Ives DG, Evans RW, Cushman M, Meilahn EN, Kuller LH. Relationship of C-reactive protein to risk of cardiovascular disease in the elderly. Results from the Cardiovascular Health Study and the Rural Health Promotion Project. Arterioscler Thromb Vasc Biol. 1997 Jun;17(6):1121-7. doi: 10.1161/01.atv.17.6.1121. PMID 9194763
- [Background] Macy EM, Hayes TE, Tracy RP. Variability in the measurement of C-reactive protein in healthy subjects: implications for reference intervals and epidemiological applications. Clin Chem. 1997 Jan;43(1):52-8. PMID 8990222
- [Background] Calles-Escandon J, Ballor D, Harvey-Berino J, Ades P, Tracy R, Sobel B. Amelioration of the inhibition of fibrinolysis in elderly, obese subjects by moderate energy intake restriction. Am J Clin Nutr. 1996 Jul;64(1):7-11. doi: 10.1093/ajcn/64.1.7. PMID 8669417
- [Background] Gubler DJ, Trent DW. Emergence of epidemic dengue/dengue hemorrhagic fever as a public health problem in the Americas. Infect Agents Dis. 1993 Dec;2(6):383-93. PMID 8012739
- [Background] Cushman M, Meilahn EN, Psaty BM, Kuller LH, Dobs AS, Tracy RP. Hormone replacement therapy, inflammation, and hemostasis in elderly women. Arterioscler Thromb Vasc Biol. 1999 Apr;19(4):893-9. doi: 10.1161/01.atv.19.4.893. PMID 10195915
- [Background] Cushman M, Lemaitre RN, Kuller LH, Psaty BM, Macy EM, Sharrett AR, Tracy RP. Fibrinolytic activation markers predict myocardial infarction in the elderly. The Cardiovascular Health Study. Arterioscler Thromb Vasc Biol. 1999 Mar;19(3):493-8. doi: 10.1161/01.atv.19.3.493. PMID 10073948
- [Background] Sakkinen PA, Macy EM, Callas PW, Cornell ES, Hayes TE, Kuller LH, Tracy RP. Analytical and biologic variability in measures of hemostasis, fibrinolysis, and inflammation: assessment and implications for epidemiology. Am J Epidemiol. 1999 Feb 1;149(3):261-7. doi: 10.1093/oxfordjournals.aje.a009801. PMID 9927222
- [Background] Smiles AM, Macy EM, Sakkinen PA, Bovill EG, Mann KG, Tracy RP. Variability in plasma prothrombin concentration: implications for use in epidemiology. Blood Coagul Fibrinolysis. 1998 Sep;9(6):525-31. doi: 10.1097/00001721-199809000-00010. PMID 9819003
- [Background] Moyer MP, Tracy RP, Tracy PB, van't Veer C, Sparks CE, Mann KG. Plasma lipoproteins support prothrombinase and other procoagulant enzymatic complexes. Arterioscler Thromb Vasc Biol. 1998 Mar;18(3):458-65. doi: 10.1161/01.atv.18.3.458. PMID 9514415
- [Background] Tracy RP. Inflammation markers and coronary heart disease. Curr Opin Lipidol. 1999 Oct;10(5):435-41. doi: 10.1097/00041433-199910000-00008. PMID 10554706
- [Background] Geffken DF, Cushman M, Burke GL, Polak JF, Sakkinen PA, Tracy RP. Association between physical activity and markers of inflammation in a healthy elderly population. Am J Epidemiol. 2001 Feb 1;153(3):242-50. doi: 10.1093/aje/153.3.242. PMID 11157411
- [Background] Lewis MR, Callas PW, Jenny NS, Tracy RP. Longitudinal stability of coagulation, fibrinolysis, and inflammation factors in stored plasma samples. Thromb Haemost. 2001 Dec;86(6):1495-500. PMID 11776319
- [Background] Burke AP, Tracy RP, Kolodgie F, Malcom GT, Zieske A, Kutys R, Pestaner J, Smialek J, Virmani R. Elevated C-reactive protein values and atherosclerosis in sudden coronary death: association with different pathologies. Circulation. 2002 Apr 30;105(17):2019-23. doi: 10.1161/01.cir.0000015507.29953.38. PMID 11980679
- [Background] Curb JD, Abbott RD, Rodriguez BL, Sakkinen P, Popper JS, Yano K, Tracy RP. C-reactive protein and the future risk of thromboembolic stroke in healthy men. Circulation. 2003 Apr 22;107(15):2016-20. doi: 10.1161/01.CIR.0000065228.20100.F7. Epub 2003 Apr 7. PMID 12681999
- [Background] Jenny NS, Tracy RP, Ogg MS, Luong le A, Kuller LH, Arnold AM, Sharrett AR, Humphries SE. In the elderly, interleukin-6 plasma levels and the -174G>C polymorphism are associated with the development of cardiovascular disease. Arterioscler Thromb Vasc Biol. 2002 Dec 1;22(12):2066-71. doi: 10.1161/01.atv.0000040224.49362.60. PMID 12482836
- [Background] Smiles AM, Jenny NS, Tang Z, Arnold A, Cushman M, Tracy RP. No association of plasma prothrombin concentration or the G20210A mutation with incident cardiovascular disease: results from the Cardiovascular Health Study. Thromb Haemost. 2002 Apr;87(4):614-21. PMID 12008943
- [Background] Sakkinen P, Abbott RD, Curb JD, Rodriguez BL, Yano K, Tracy RP. C-reactive protein and myocardial infarction. J Clin Epidemiol. 2002 May;55(5):445-51. doi: 10.1016/s0895-4356(01)00502-9. PMID 12007546
- [Background] Liu Y, Coresh J, Eustace JA, Longenecker JC, Jaar B, Fink NE, Tracy RP, Powe NR, Klag MJ. Association between cholesterol level and mortality in dialysis patients: role of inflammation and malnutrition. JAMA. 2004 Jan 28;291(4):451-9. doi: 10.1001/jama.291.4.451. PMID 14747502
- [Background] Tracy RP. Thrombin, inflammation, and cardiovascular disease: an epidemiologic perspective. Chest. 2003 Sep;124(3 Suppl):49S-57S. doi: 10.1378/chest.124.3_suppl.49s. PMID 12970124